CLINICAL TRIAL: NCT02512874
Title: Does Pulmonary Rehabilitation Improve Frailty in Chronic Lung Disease?
Brief Title: Does Pulmonary Rehabilitation Improve Frailty?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Cassie C. Kennedy, M.D., Consultant for Critical Care Medicine, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15-001230; K23HL128859 (NIH)
Record Dates: First submitted 2015-07-24; First posted 2015-07-31 (Estimated); Results first posted 2018-10-05 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Disease, Pulmonary
MeSH Terms: conditions — Lung Diseases | interventions — Muscle Strength Dynamometer; Fitness Trackers; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Pulmonary Rehabilitation (Other): One arm study - all participants will go to pulmonary rehabilitation, received questionnaires, Dual-energy X-ray absorptiometry (DEXA) scans, Dynamometer and gait speed tests and activity measured through an activity monitor.
  Interventions: Other: Pulmonary Rehabilitation; Device: Dynamometer; Radiation: DEXA; Other: Gait Speed Test; Device: Activity Monitor; Other: Questionnaires

INTERVENTIONS:
Other: Pulmonary Rehabilitation — Measures of frailty taken before and after pulmonary rehabilitation.
Device: Dynamometer — Grip Test
Radiation: DEXA — Body Composition Testing
Other: Gait Speed Test — 15 foot walk test
Device: Activity Monitor — Measures energy expenditure and activity
Other: Questionnaires — Health-related questionnaires measuring self-reported exhaustion, emotions and disease symptoms.

SUMMARY:
Frailty is a state of health with predisposition to adverse events, morbidity and mortality. Frailty consists of weakness, slowness, low physical activity, exhaustion, and wasting. Frailty is associated with increased hospitalizations and death in lung disease. It is unknown if pulmonary rehabilitation will improve frailty markers.

DETAILED DESCRIPTION:
Individuals referred to pulmonary rehabilitation will be examined for frailty markers. After completing pulmonary rehabilitation, the same tests will be performed. The effects of pulmonary rehabilitation will be examined.

ELIGIBILITY:
Inclusion criteria:

* Referred for pulmonary rehabilitation
* consenting to research

Exclusion criteria:

-Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-07-21; Primary Completion 2018-10-16 (Actual); Study Completion 2018-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cassie Kennedy, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Pulmonary Rehabilitation: One arm study - all participants will go to pulmonary rehabilitation, received questionnaires, DEXA scans, Dynamometer and gait speed tests and activity measured through an activity monitor.
  Pulmonary Rehabilitation: Measures of frailty taken before and after pulmonary rehabilitation.
  Dynamometer: Grip Test
  DEXA: Body Composition Testing
  Gait Speed Test: 15 foot walk test
  Activity Monitor: Measures energy expenditure and activity
  Questionnaires: Health-related questionnaires measuring self-reported exhaustion, emotions and disease symptoms.
Period: Overall Study
Arm/Group | Pulmonary Rehabilitation
Started | 65
Completed | 63
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Pulmonary Rehabilitation
Number analyzed (Participants) | 63
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65 [59.0 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 54
  More than one race | 0
  Unknown or Not Reported | 9
Region of Enrollment [Number; unit: participants]
  United States | 63
Primary Pulmonary Diagnosis [Count of Participants; unit: Participants]
  Obstructive | 35
  Post Lung Transplant | 13
  Interstitial Lung Disease | 10
  Other | 5
Pulmonary Function - Forced expiratory volume [Median (Inter-Quartile Range); unit: liters] — The forced expiratory volume in one second (FEV1) measurement shows the amount of air in liters a person can forcefully exhale in one second.
  liters | 1.3 [1.0 to 2.0]
Pulmonary Function - % Predicted [Median (Inter-Quartile Range); unit: percent] — The % predicted represents the percent of the lung size that can be exhaled in one second.
  percent | 49 [39 to 66]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Frailty Phenotype at Baseline and 6 Months
Description: Frailty phenotype is 3 or more of: slow gait speed, exhaustion, decreased hand grip strength, decreased activity level, or wasting. Grip strength parameters, gait speed, exhaustion per Fried et al. 2001. Wasting is defined as further decrease in fat free mass by body composition measurement using DEXA. Low physical activity would be activity monitor in lower quartile.
Time Frame: Baseline, Six months
Population: Forty-nine participants (77.8%) of the 63 participants completed at lease one follow-up frailty parameter assessment after completion of pulmonary rehabilitation.
Measure: Count of Participants; unit: Participants
Arm/Group | Pulmonary Rehabilitation
Number analyzed (Participants) | 63
Participants
  Baseline | 24
  Six months: number analyzed (Participants) | 49
  Six months | 15
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation; Test type: Superiority; p = 0.62, Chi-squared

2. Secondary Outcome: Wasting
Description: DXA measurement of body mass index pre- and post- PR.
Time Frame: after pulmonary rehabilation completion, appoximately 8 weeks
Population: Data for 37 participants was available for analysis.
Measure: Median (Inter-Quartile Range); unit: kg/m^2
Arm/Group | Pulmonary Rehabilitation
Number analyzed (Participants) | 37
kg/m^2 | 0.04 [-0.4 to 1.1]

3. Secondary Outcome: Change in Strength
Description: Change in Grip Strength as measured by hand dynamometer.
Time Frame: after completion of pulmonary rehab, approximately 8 weeks
Population: Data for 45 participants was available for analysis.
Measure: Median (Inter-Quartile Range); unit: kg
Arm/Group | Pulmonary Rehabilitation
Number analyzed (Participants) | 45
kg | 0 [-1.6 to 2.6]

4. Secondary Outcome: Change in Gait Speed
Description: gait speed test measured over 15 feet
Time Frame: pre and post pulmonary rehab, approximately 8 weeks
Population: Data for 43 participants was available for analysis.
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Pulmonary Rehabilitation
Number analyzed (Participants) | 43
seconds | -0.6 [-1.5 to 0.5]

5. Secondary Outcome: Improvement in Exhaustion
Description: Self-reported exhaustion - measured by two questions in the Center for the Epidemiological Studies in Depression (CES-D) scale and reported as a dichotomous variable (exhausted or not exhausted).
Time Frame: pre and post pulmonary rehab, approximately 8 weeks
Population: Data for 39 participants was available for analysis. 19 participants were exhausted pre-pulmonary rehabilitation. 17 were exhausted following pulmonary rehab.
Measure: Count of Participants; unit: Participants
Arm/Group | Pulmonary Rehabilitation
Number analyzed (Participants) | 39
Participants | 2

6. Secondary Outcome: Change in Physical Activity Level
Description: Measured by Body Media armband activity monitor using total energy expenditure divided by the resting metabolic rate
Time Frame: pre and post pulmonary rehab, approximately 8 weeks
Population: Data for 47 participants was available for analysis.
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Pulmonary Rehabilitation
Number analyzed (Participants) | 47
ratio | 0.4 [-0.4 to 1.1]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from baseline through 6 month follow up.
Arm/Group | Pulmonary Rehabilitation
All-Cause Mortality (participants affected / at risk) | 4/65
Serious Adverse Events (participants affected / at risk) | 0/65
Other Adverse Events (participants affected / at risk) | 0/65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-23): https://cdn.clinicaltrials.gov/large-docs/74/NCT02512874/Prot_SAP_000.pdf